CLINICAL TRIAL: NCT02080117
Title: Adequate Definition of Delayed Graft Function in Living and Deceased Donor Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, WonHo Kim, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-12-089
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Deceased Donor Kidney Transplantation; Living Donor Kidney Transplantation
Keywords: kidney transplantation; delayed graft function; creatinine; graft survival
MeSH Terms: conditions — Delayed Graft Function | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients who underwent kidney transplantation: patients who underwent living or deceased donor kidney transplantation between 2008 and 2013
  Interventions: Procedure: kidney transplantation, living or deceased donor

INTERVENTIONS:
Procedure: kidney transplantation, living or deceased donor

SUMMARY:
It is required to establish an adequate definition of delayed graft function in deceased donor kidney transplantation. We attempt to compare various definitions of delayed graft function and find the definition that can predict graft function survival best in deceased donor kidney transplantation.

DETAILED DESCRIPTION:
Delayed graft function after kidney transplantation has been reported to be an important predictor for poor short and long-term survival. Delayed graft function increases post-transplantation morbidity, hospital stay, and incidence of premature graft failure. However, the definition of delayed graft function varies and more than ten definitions have been used in previous studies. Although the definition using dialysis requirements during seven days after transplantation has been used most frequently, dialysis may be required without any evidence of renal damage during one week after transplantation. Furthermore, the incidence of delayed graft function in living donor kidney transplantation using this definition has been reported to be relatively low (as low as 1.6%) compared with the incidence in deceased donor kidney transplantation (up to 50%). Therefore, it is required to establish a better definition of delayed graft function in deceased donor kidney transplantation. We attempt to compare various definitions of delayed graft function in deceased donor kidney transplantation and find the definition that can predict graft function survival best in deceased donor kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent living or deceased donor kidney transplantation between 2008 and 2013

Exclusion Criteria:

* incomplete data of postoperative creatinine during ten days after transplantation or postoperative urine output during three days after transplantation
* patients who underwent retransplantation
* patients who expired for reasons other than kidney transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent living or deceased donor kidney transplantation between 2008 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
delayed graft function as defined by dialysis requirements within one week after transplantation | during 7 days after transplantation
  delayed graft function as defined by dialysis requirements within one week after transplantation

SECONDARY OUTCOMES:
delayed graft function as defined by urine output less than1200 ml during first day after transplantation | during 24 hours after transplantation
  delayed graft function as defined by urine output less than1200 ml during first day after transplantation
delayed graft function as defined by serum creatinine decrease less than 10% during 48 hours after transplantation | during 48 hours after transplantation
  delayed graft function as defined by serum creatinine decrease less than 10% during 48 hours after transplantation
delayed graft function as defined by creatinine greater than 2.5 mg/dL at ten days after transplantation | after ten days after transplantation
  delayed graft function as defined by creatinine greater than 2.5 mg/dL at ten days after transplantation
delayed graft function as defined by creatinine clearance less than 10 ml/min/1.73m2 during 24 hours after transplantation | during 24 hours after transplantation
  delayed graft function as defined by creatinine clearance less than 10 ml/min/1.73m2 during 24 hours after transplantation
delayed graft function as defined by creatinine did not decrease less than preoperative value | during one week after transplantation
  delayed graft function as defined by creatinine did not decrease less than preoperative value

OTHER OUTCOMES:
graft survival | one month, six month, and one year after transplantation
  graft survival one month, six month, and one year after transplantation
Mortality | one month, six month, and one year after transplantation
  Mortality after one month, six month, and one year after transplantation
immediate graft function | after eight days after transplantation
  immediate graft function after eight days after transplantation (defined as serum creatinine decrease less than 70% of preoperative value)
slow graft function | at eight days after transplantation
  slow graft function at eight days after transplantation (defined as serum creatinine greater than 70% of preoperative value)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea